CLINICAL TRIAL: NCT02568150
Title: Single Arm, Open, Single Institute, Domestic Phase 4 Clinical Study to Evaluate the Onset Time of Improvement of Glabellar Frown Lines and Safety of DWP450-004 Injection for Adults With Worse Than Moderate Glabellar Frown Lines
Brief Title: Evaluation Onset Time of DWP450-004 and Safety in Moderate-severe Glabellar Lines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP450004
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Moderate-severe Glabellar Lines
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): Onset time of improvement effect of glabellar lines at maximum frown of botulinum toxin treatment
  Interventions: Biological: Single group, open-label

INTERVENTIONS:
Biological: Single group, open-label

SUMMARY:
Evaluate onset time and safety of improvement effect of each group's forehead wrinkles after 2, 3, 4, 5, 14 days from administration of 20U dosage of DWP450-004 for adult patients who need more than moderate improvement of forehead wrinkles.

DETAILED DESCRIPTION:
Currently, botulinum type A toxin related products are used not only in treatment areas but they are used often in cosmetic area as well and frequency of usage is increasing as well. Daewoong Pharmaceutical Co., Ltd. has developed a safe product by identifying wild-type Clostridium botulinum (type A) strain and purifying high purity, high quality botulinum toxin type A proteins from the strain. As a result of characteristic analysis (genotype analysis, morphological / biochemical characteristic verification test, toxicity test, etc) of the identified fungi, it was confirmed that the biological and chemicophysical properties are equal to those of wild-type Clostridium botulinum (type A, Hall strain).

Regarding treatment satisfaction of those patients who were administered with botulinum toxin product, onset time plays an important role as a factor. Limitation found when reviewing the existing publications was in defining onset time solely on the determination of effect simply on response to whether there was an improvement. However, this study defines improvement rate of glabellar lines as ratio of reduction of more than 1 point from the baseline by investigator and thus it appears more objective data can be obtained than existing studies. Therefore, with this background, we intend to conduct phase 4 clinical study to explore onset time for DWP450-004 injection's glabellar lines improvement effect.

ELIGIBILITY:
Inclusion Criteria

1. Males and Females who are at least 20 years old and not older than 65 years old
2. Subjects who have a least 2 points (moderate) of glabellar lines at maximum frown to the maximum confirmed with investigator's line assessment severity.
3. Subjects who can comply well with clinical study procedures and visit schedules
4. Subjects who voluntarily signed the Informed Consent Form

Exclusion Criteria

1. Subjects with diseases that can affect neuromuscular functioning such as oderate muscle weakness, Eaton-Lambert Syndrome, Amyotrophic side sclerosis, motor neuropathy, etc.
2. Subjects who took aminoglycoside antibiotics, curare-like agents or drugs that inhibit neuromuscular functioning (including muscle relaxants, anticholinergic type, benzodiazepine type, benzamide type, tetracycline type, or lincomycin type of antibiotics) within 4 weeks prior to screening
3. Subjects with skin abnormality near the injection site such as infection, skin disease, or scar
4. In case where subject underwent other procedures that may affect the glabellar lines or brow area within 6 months prior to screening
5. Subjects who received botulinum Type A toxin products within 8 months prior to screening or received botulinum Type B products within 8 months prior to screening
6. Subjects whose glabellar lines cannot be satisfactorily improved with physical method since the lines are not flattened even using hands.
7. Subjects with facial paralysis or history of blepharoptosis
8. Subjects who are pregnant, lactating or who plan to be pregnant during the clinical period or females of child bearing years who do not use available contraceptive methods (subjects of child bearing years must be negative from a pregnancy test prior to injection.)
9. Subjects allergic to or sensitive to the Investigational Product or applicable ingredients
10. Subjects taking aspirin, NSAIDs or anticoagulant
11. Subjects who have participated in another clinical study within 30 days prior to screening or patient who participated in a clinical study and the period of 5 times the Investigational Product's half life has not passed
12. Other subjects who are deemed not to be appropriate for this clinical study in the discretion of investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Onset time of improvement effect of glabellar lines at maximum frown confirmed with Investigator's line assessment severity after administration | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Joon Pio Hong, MD, Study Chair — Asan Medical Center